CLINICAL TRIAL: NCT06832241
Title: ÉVALUATION DE LA CHARGE COGNITIVE DES PILOTES D'HÉLICOPTÈRES EN FORMATION "ECCOLicoF"
Brief Title: Cognitive Load Assessment of Helicopter Pilots in Training
Acronym: ECCOLicoF
Status: Not yet recruiting | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2023PBMD04; 2024-A01855-42 (Other: IDRCB)
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Cognitive Impairment; Situational Anxiety; Skills, Coping
Keywords: Cognitive load; Military helicopter pilots
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to identify the effect of the increase of the situation demands, with or without a thread, on military helicopter pilot's cognitive load, depending on their skills acquisition (at the beginning, midway and end of training course). This study is carried out on a simulator, in virtual reality and allows to identify the moments of cognitive load enhancement and the associated indicators such as subjective, physiological and behavioural indicators. Recommendations will be done to go towards an individualization of the lessons during the pilots education, by anticipating an overload which has a deleterious effect on learning.

ELIGIBILITY:
Inclusion Criteria:

* Being a trainee at the Instructional center of helicopter crews
* Being more than 18 years old
* Being insured under the French social security system
* Having the bases to pilot helicopters
* Having signed the non-opposition form

Exclusion Criteria:

* Being minor or an incapacitated adult
* Being in a motor handicap situation
* Having a cardiac pathology
* Having a visual pathology that is uncorrected by glasses or lens
* Having a bad audition
* Having a psychiatric disorder, a neurologic or organic disorder requiring a medical treatment
* Taking psychotropics
* Drinking more than 28 units of alcohol per week
* Being epileptic

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Military helicopter pilots trainees
Sampling Method: Non-Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Subjective level of cognitive load | It is completed during 5 minutes after each of the six scenarios
  The NASA-TLX questionnaire is used to assess the subjective level of cognitive load

SECONDARY OUTCOMES:
Objective level of cognitive load | It is measured during each of the six scenarios lasting around 5 minutes
  It is measures by physiological indicators ( cardiac activity and electroencephalogram) and behavioural indicators (tasks performance, ocular saccades and blinks)
Subjective level of anxiety | It is measured during 1 minute after each of the six scenarios
  It is measured by a visual analogue scale
Objective level of anxiety | It is measured during each of the six scenarios lasting around 5 minutes
  It is measured by the electrodermal activity
Subjective level of fatigue | It is measured during 1 minute before each of the six scenarios
  It is measured by the Karolinska Sleepiness Scale

CONTACTS AND LOCATIONS:
Overall Officials: Julie ALBENTOSA, Study Chair — IRBA, 1 place Valérie André, 91 223 Brétigny-sur-Orge cedex